CLINICAL TRIAL: NCT00414973
Title: Comparison of Teriparatide and Calcitonin in the Treatment of Men and Postmenopausal Women With Osteoporosis
Brief Title: A Study for Patients With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10591; B3D-MC-GHDG
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; salmon calcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Teriparatide
- B (Active Comparator)
  Interventions: Drug: Salmon Calcitonin

INTERVENTIONS:
Drug: Teriparatide — Subcutaneous, 20 micrograms/day, 24 weeks
  Other Names: LY333334; Forteo; Forsteo
  Arms: A
Drug: Salmon Calcitonin — Intranasal, 200 International Units (IU)/day, 24 weeks
  Arms: B

SUMMARY:
The purpose of this study is to compare the effect of injectable teriparatide to intranasal salmon calcitonin on lumbar spine bone mineral density, in the treatment of Chinese patients with established osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoporosis
* No other severe disabling conditions
* Should have at least 1 vertebral or non-vertebral prevalent fracture, and bone mineral density T-score should be less than -2.5
* Ambulatory
* Men (aged 40 to 85 years) or postmenopausal women (aged 55 to 85 years)

Exclusion Criteria:

* History of a disease that affects bone metabolism
* History of treatment with any drug that may significantly affect bone metabolism
* History or presence of liver disease
* History or presence of kidney disease
* History of excessive alcohol drinking or drug abuse

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- China (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenzhou

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 364 participants were randomized, but 2 females did not receive study drug and are not included in any of the analyses.
Groups:
- Teriparatide - Females; Teriparatide - Males: Subcutaneous, 20 micrograms/day, 24 weeks
- Calcitonin - Females: Intranasal, 200 International Units (IU)/day, 24 weeks
- Calcitonin - Males: Intranasal, 200 IU/day, 24 weeks
Period: Overall Study
Arm/Group | Teriparatide - Females | Calcitonin - Females | Teriparatide - Males | Calcitonin - Males
Started | 218 | 109 | 24 | 11
Completed | 190 | 99 | 21 | 11
Not Completed | 28 | 10 | 3 | 0
Not completed — Withdrawal by Subject | 14 | 4 | 1 | 0
Not completed — Adverse Event | 10 | 0 | 1 | 0
Not completed — Protocol Violation | 3 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide - Females | Calcitonin - Females | Teriparatide - Males | Calcitonin - Males | Total
Number analyzed (Participants) | 218 | 109 | 24 | 11 | 362
Age Continuous [Mean (Standard Deviation); unit: years] | 69.09 (6.95) | 67.81 (7.22) | 68.27 (8.28) | 67.39 (11.01) | 68.60 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 109 | 0 | 0 | 327
  Male | 0 | 0 | 24 | 11 | 35
Region of Enrollment [Number; unit: participants]
  China | 218 | 109 | 24 | 11 | 362
Race/Ethnicity [Number; unit: participants]
  East Asian | 218 | 109 | 24 | 11 | 362
Duration of Osteoporosis [Mean (Standard Deviation); unit: years] | 3.6 (5.33) | 3.1 (4.16) | 1.9 (2.24) | 2.4 (2.54) | 3.30 (4.80)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline to 24 Week Endpoint in Lumbar Spine Bone Mineral Density (BMD), Postmenopausal Women
Description: Lumbar spine bone mineral density (milligrams per square centimeter) was measured by dual energy X-ray absorptiometry (DXA). Change = Endpoint minus baseline.
Time Frame: Baseline to 24 weeks
Population: Number of Intention to Treat patients with baseline and at least one post baseline measurement. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: percentage change in lumbar spine BMD
Groups:
- Calcitonin - Females: Intranasal, 200 IU/day, 24 weeks
Arm/Group | Teriparatide - Females | Calcitonin - Females
Number analyzed (Participants) | 201 | 102
percentage change in lumbar spine BMD | 6.04 (0.48) | 1.65 (0.65)
Statistical Analysis 1: Comparison: Teriparatide - Females vs Calcitonin - Females; Null hypothesis=no difference between percentage changes from baseline in lumbar spine bone mineral density for female patients receiving teriparatide compared to female patients receiving calcitonin; Test type: Superiority or Other; p < 0.0001, ANCOVA — There were no adjustments for multiple comparisons; Mean Difference (Net) = 4.39, 95% CI [2.89 to 5.89], Standard Error of Mean 0.76 — Difference = Teriparatide minus Calcitonin

2. Secondary Outcome: Percentage Change From Baseline to 24 Week Endpoint in Total Hip Bone Mineral Density (BMD), Postmenopausal Women
Description: Total hip bone mineral density (milligrams per square centimeter) was measured by dual energy X-ray absorptiometry (DXA). Change = Endpoint minus baseline.
Time Frame: Baseline to 24 weeks
Population: Number of Intention to Treat patients with baseline plus at least one post baseline measurement. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: percentage change in total hip BMD
Arm/Group | Teriparatide - Females | Calcitonin - Females
Number analyzed (Participants) | 205 | 104
percentage change in total hip BMD | -0.53 (0.44) | -0.62 (0.59)
Statistical Analysis 1: Comparison: Teriparatide - Females vs Calcitonin - Females; Test type: Superiority or Other; p = 0.9062, ANCOVA; Mean Difference (Net) = 0.08, 95% CI [-1.30 to 1.46], Standard Error of Mean 0.70 — Difference = Teriparatide minus Calcitonin

3. Secondary Outcome: Percentage Change From Baseline to 12 Weeks and 24 Weeks in Osteocalcin, Postmenopausal Women
Description: Measures of serum osteocalcin (nanograms per milliliter). Change = Endpoint minus baseline.
Time Frame: Baseline to 12 weeks and 24 weeks
Population: Number of Intention to Treat patients with measurements at respective visits.
Measure: Median (Inter-Quartile Range); unit: percentage change in osteocalcin
Arm/Group | Teriparatide - Females | Calcitonin - Females
Number analyzed (Participants) | 218 | 109
percentage change in osteocalcin
  Week 12 Percentage Change (n=202, n=102) | 113.87 (21.46) [61.20 to 175.94] | -7.67 (5.43) [-20.51 to 12.56]
  Week 24 Percentage Change (n=191, n=97) | 137.45 (36.53) [74.34 to 261.68] | -10.58 (8.21) [-25.69 to 7.33]
Statistical Analysis 1: Comparison: Teriparatide - Females vs Calcitonin - Females; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank-Sum Test — P-value for Week 12 Percentage Change
Statistical Analysis 2: Comparison: Teriparatide - Females vs Calcitonin - Females; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank-Sum Test — P-value for Week 24 Percentage Change

4. Secondary Outcome: Percentage Change From Baseline to 24 Week Endpoint in Lumbar Spine Bone Mineral Density (BMD), Men
Description: as for outcome 1
Time Frame: Baseline to 24 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change in lumbar spine BMD
Arm/Group | Teriparatide - Males | Calcitonin - Males
Number analyzed (Participants) | 21 | 10
percentage change in lumbar spine BMD | 6.01 (1.20) | 3.38 (1.77)
Statistical Analysis 1: Comparison: Teriparatide - Males vs Calcitonin - Males; Test type: Superiority or Other; p = 0.2409, ANCOVA; Mean Difference (Net) = 2.63, 95% CI [-1.87 to 7.13], Standard Error of Mean 2.20 — Difference = Teriparatide minus Calcitonin

5. Secondary Outcome: Percentage Change From Baseline to 24 Week Endpoint in Total Hip Bone Mineral Density (BMD), Men
Description: as for outcome 2
Time Frame: Baseline to 24 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change in total hip BMD
Arm/Group | Teriparatide - Males | Calcitonin - Males
Number analyzed (Participants) | 21 | 11
percentage change in total hip BMD | 0.37 (1.11) | 1.34 (1.54)
Statistical Analysis 1: Comparison: Teriparatide - Males vs Calcitonin - Males; Test type: Superiority or Other; p = 0.6156, ANCOVA; Mean Difference (Net) = -0.96, 95% CI [-4.85 to 2.92], Standard Error of Mean 1.90 — Difference = Teriparatide minus Calcitonin

6. Secondary Outcome: Percentage Change From Baseline to 12 Weeks and 24 Weeks in Osteocalcin, Men
Description: Measures of serum osteocalcin (nanograms per milliliter). Change = Endpoint minus baseline.
Time Frame: Baseline to 12 weeks and 24 weeks
Population: Number of Intention to Treat patients with measurements at respective visit.
Measure: Median (Inter-Quartile Range); unit: percentage change in osteocalcin
Arm/Group | Teriparatide - Males | Calcitonin - Males
Number analyzed (Participants) | 24 | 11
percentage change in osteocalcin
  Week 12 Percentage Change (n=21, n=11) | 107.27 (14.88) [45.16 to 181.85] | 4.35 (13.48) [-15.83 to 18.95]
  Week 24 Percentage Change (n=21, n=11) | 79.26 (26.94) [13.06 to 142.86] | -17.65 (5.21) [-27.95 to 3.08]
Statistical Analysis 1: Comparison: Teriparatide - Males vs Calcitonin - Males; Test type: Superiority or Other; p = 0.0026, Wilcoxon Rank-Sum Test — P-value for Week 12 Percentage Change
Statistical Analysis 2: Comparison: Teriparatide - Males vs Calcitonin - Males; Test type: Superiority or Other; p = 0.0006, Wilcoxon Rank-Sum Test — P-value for 24 Week Percentage Change

ADVERSE EVENTS:
Arm/Group | Teriparatide - Females | Calcitonin - Females | Teriparatide - Males | Calcitonin - Males
Serious Adverse Events (participants affected / at risk) | 8 | 1 | 2 | 0
Other Adverse Events (participants affected / at risk) | 67 | 26 | 7 | 0
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Teriparatide - Females | Calcitonin - Females | Teriparatide - Males | Calcitonin - Males
Acute myocardial infarction (Cardiac disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Angina pectoris (Cardiac disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Atrial fibrillation (Cardiac disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Cardiac discomfort (Cardiac disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Cardiac disorder (Cardiac disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Heart valve incompetence (Cardiac disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Multi-organ failure (General disorders) | 0/217 (0) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Pneumonia (Infections and infestations) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Sinusitis fungal (Infections and infestations) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/217 (0) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Cerebral infarction (Nervous system disorders) | 0/217 (0) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/217 (0) | 1/110 (1) | 0/24 (0) | 0/11 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0/217 (0) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Arteriosclerosis obliterans (Vascular disorders) | 1/217 (1) | 0/110 (0) | 0/24 (0) | 0/11 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Teriparatide - Females | Calcitonin - Females | Teriparatide - Males | Calcitonin - Males
Palpitations (Cardiac disorders) | 6/217 (8) | 1/110 (1) | 0/24 (0) | 0/11 (0)
Diarrhoea (Gastrointestinal disorders) | 2/217 (2) | 2/110 (3) | 1/24 (1) | 0/11 (0)
Nausea (Gastrointestinal disorders) | 11/217 (15) | 0/110 (0) | 0/24 (0) | 0/11 (0)
Asthenia (General disorders) | 3/217 (3) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Thirst (General disorders) | 1/217 (1) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Nasopharyngitis (Infections and infestations) | 7/217 (7) | 4/110 (5) | 1/24 (1) | 0/11 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0/217 (0) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Alanine aminotransferase increased (Investigations) | 0/217 (0) | 1/110 (1) | 1/24 (1) | 0/11 (0)
Aspartate aminotransferase increased (Investigations) | 0/217 (0) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Blood alkaline phosphatase increased (Investigations) | 10/217 (10) | 1/110 (1) | 1/24 (1) | 0/11 (0)
Blood creatine phosphokinase increased (Investigations) | 2/217 (2) | 1/110 (1) | 1/24 (1) | 0/11 (0)
Blood uric acid increased (Investigations) | 10/217 (10) | 0/110 (0) | 1/24 (1) | 0/11 (0)
Gamma-glutamyltransferase increased (Investigations) | 1/217 (1) | 1/110 (1) | 1/24 (1) | 0/11 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6/217 (8) | 1/110 (3) | 0/24 (0) | 0/11 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12/217 (19) | 4/110 (8) | 0/24 (0) | 0/11 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10/217 (19) | 2/110 (3) | 1/24 (1) | 0/11 (0)
Dizziness (Nervous system disorders) | 16/217 (23) | 4/110 (5) | 2/24 (2) | 0/11 (0)
Headache (Nervous system disorders) | 5/217 (7) | 4/110 (6) | 0/24 (0) | 0/11 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days